CLINICAL TRIAL: NCT01810770
Title: A Single-arm, International, Prospective, Interventional, Open-label, Multicenter Study of Radium-223 Dichloride in the Treatment of Patients With Castration-Resistant Prostate Cancer (CRPC) With Bone Metastasis.
Brief Title: Radium-223 Dichloride Asian Population Study in the Treatment of CRPC Patients With Bone Metastasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15397
Record Dates: First submitted 2013-03-12; First posted 2013-03-14 (Estimated); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Prostatic Neoplasms
Keywords: Radium-223 Dichloride; Prostatic Neoplasms; Bone Metastasis
MeSH Terms: conditions — Prostatic Neoplasms | interventions — radium Ra 223 dichloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radium-223 dichloride (Experimental)
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY88-8223)

INTERVENTIONS:
Drug: Radium-223 dichloride (Xofigo, BAY88-8223) — Radium-223 dichloride, 55 kBq/kg body weight, will be administered as a slow bolus IV injection at 4 week intervals for up to 6 doses.

SUMMARY:
To evaluate the safety and efficacy (Overall survival [OS]) of multiple doses of Ra-223 dichloride in an Asian population of subjects with CRPC metastatic to the bone.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate
* Patients diagnosed with progressive bone predominant metastatic Castration-Resistant Prostate Cancer (CRPC) /Hormone Refractory Prostate Cancer (HRPC) with at least 2 skeletal metastases on imaging with no lung, liver, and/or brain metastasis (lymph node only metastasis is allowed)
* Known hormone refractory disease
* No intention to use cytotoxic chemotherapy within the next 6 months
* Either regular (not occasional) analgesic medication use for cancer related bone pain or treatment with external bean radiation therapy (EBRT) for bone pain within previous 12 weeks
* Age >/= 18 years
* Race is Asian
* Eastern Co-operative Oncology Group (ECOG) Performance Status (PS): 0-2
* Life expectancy >/= 6 months
* Adequate bone marrow, liver and renal function as assessed by the Laboratory required by protocol

Exclusion Criteria:

* Treatment with an investigational drug within previous 4 weeks prior to screening, or planned during the treatment or follow-up periods
* Eligible for docetaxel treatment, i.e. subjects who are fit enough, willing and who are located where treatment with docetaxel is available
* Treatment with cytotoxic chemotherapy within previous 4 weeks prior to screening, or failure to recover from adverse events due to cytotoxic chemotherapy administered more than 4 weeks prior to screening (however ongoing neuropathy is permitted)
* Prior hemibody external radiotherapy is excluded. Subjects who received other types of prior external radiotherapy are allowed provided that the bone marrow function is assessed and meets the protocol requirements for hemoglobin, absolute neutrophil count and platelets.
* Received systemic therapy radionuclides (e.g., strontium-89, samarium-153, rhenium-186, rhenium-188, or radium-223 dichloride) for the treatment of bony metastases
* Blood transfusion or erythropoetin stimulating agents within the previous 4 weeks prior to screening
* Other malignancy treated within the last 3 years (except non-melanoma skin cancer or low-grade superficial bladder cancer)
* Visceral metastases as assessed by abdominal/pelvic computed tomography (CT) or other imaging modality
* Presence of brain metastases
* Lymphadenopathy exceeding 3 cm in short-axis diameter
* Any size pelvic lymphadenopathy if it is thought to be a contributor to concurrent hydronephrosis
* Imminent or established spinal cord compression based on clinical findings and/or magnetic resonance imaging (MRI). Subjects with history of spinal cord compression should have completely recovered.
* Received local practice implant therapy containing lodine-125 or Palladium-103 for the primary lesion of prostate cancer within the 6 months prior to screening.
* Any other serious illness or medical condition

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2013-03-26 (Actual); Primary Completion 2017-09-25 (Actual); Study Completion 2017-09-25 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | Up to 36 months
Number of participants with laboratory changes | Up to 36 months
Number of participants with changes in vital signs | Up to 36 months
Number of participants with changes in electrocardiogram (ECG) | Up to 36 months
Overall Survival (OS) | Up to 36 months
  OS is defined as the time from date of first study drug treatment to death due to any cause. Subjects still alive at the time of analysis were censored at their last date of last contact.

SECONDARY OUTCOMES:
Changes in total Alkaline Phosphate (ALP) in serum | Up to 36 months
Number of participants with total-ALP normalization | Up to 36 months
Time to total ALP progression | Up to 36 months
Changes in prostate specific antigen (PSA) in serum | Up to 36 months
Time to PSA progression | Up to 36 months
Time to first skeletal related event (SRE) | Up to 36 months
SRE free survival | Up to 36 months
Time to occurrence of first use of radio-isotopes to relieve skeletal symptoms | Up to 36 months
Time to occurrence of first start of any other anti-cancer treatment | Up to 36 months
Time to occurrence of first deterioration of Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) | Up to 36 months
Quality of life (QoL) | Up to 36 months
  QoL is assessed by the scores got from the Functional Assessment of Cancer Therapy in subjects with prostate cancer (FACT-P) questionnaire, EuroQoL (EQ-5D) questionnaire, and the BPI-SF questionnaire.
Time to pain progression | Up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (12):
- China (5):
  - Guangzhou, Guangdong
  - Nanjing, Jiangsu
  - Beijing
  - Guangzhou
  - Shanghai
- Singapore, Singapore
- South Korea (2):
  - Donggu, Gwangju Gwang''yeogsi
  - Seoul
- Taiwan (4):
  - Taipei City, Taipei
  - Kaohsiung City
  - Taipei
  - Taoyuan District